CLINICAL TRIAL: NCT05564884
Title: The Association of Neonatal SARS-CoV-2 Anti-spike Protein Receptor-binding Domain Antibodies at Delivery With Infant COVID-19 Infection Under Age 6 Months: a Prospective Cohort Study
Brief Title: Neonatal SARS-CoV-2 Anti-spike Protein Receptor-binding Domain Antibodies at Delivery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RMC-0275-21
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unvaccinated, Prior natural COVID-19 infection: Unvaccinated, Prior natural COVID-19 infection
  Interventions: Other: no intervantion
- Vaccinated, No prior natural COVID-19 infection: Vaccinated, No prior natural COVID-19 infection
  Interventions: Other: no intervantion
- Vaccinated, Prior natural COVID-19 infection: Vaccinated, Prior natural COVID-19 infection
  Interventions: Other: no intervantion

INTERVENTIONS:
Other: no intervantion — no intervention

SUMMARY:
To assess the association between neonatal SARS-CoV-2 antibody level at delivery and infant COVID-19 infection under age 6 months, and to identify predictive factors for neonatal antibody level at delivery.

DETAILED DESCRIPTION:
This prospective observational study was conducted at the Rabin Medical Center, Israel. Mothers were enrolled from September 2021 to mid-February 2022, prior to transfer to the delivery room, and followed at the Maternity and Infant Ward. The study was approved by the institutional ethics committee (RMC- 0275-21). Written informed consent was obtained from the participating mothers. Inclusion criteria included maternal recipient of at least one dose of the BNT162b2 mRNA COVID-19 vaccine or prior microbiologically-confirmed natural COVID-19 infection. Exclusion criteria included (a) preterm birth at <34 weeks gestation; (b) congenital or acquired immune deficiency, including recipient of biological agents during the prior year to enrolment.

ELIGIBILITY:
Inclusion Criteria:

included maternal recipient of at least one dose of the BNT162b2 mRNA COVID-19 vaccine or prior microbiologically-confirmed natural COVID-19 infection

Exclusion Criteria:

(a) preterm birth at <34 weeks gestation; (b) congenital or acquired immune deficiency, including recipient of biological agents during the prior year to enrolment.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Mothers prior to transfer to the delivery room and followed at the Maternity and Infant Ward
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2021-09-12 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
neonatal anti-spike antibody levels | 6 months
  Primary outcomes were neonatal anti-spike antibody levels at delivery and infant microbiologically-confirmed COVID-19 infection at age <6 months

CONTACTS AND LOCATIONS:
Overall Officials: Liat Ashkenazi-Hoffnung, Principal Investigator — Schneider children medical center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No
According to ethics committee approval.